CLINICAL TRIAL: NCT06520189
Title: Value of F-18 FDG PET/CT for the Prediction of EGFR Mutation in Lung Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Walaa Gamal Fathy, Assistant lecturer, Assiut University
Other Study IDs: F-18 FDG PET/CT and EGFR
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: F-18 FDGPET/CT — F-18 FDGPET/CT oncology protocol for lung cancer patients

SUMMARY:
To detect value of F-18FDG PET/CT as a non-invasive method for the prediction of EGFR mutations in lung cancer patients.

DETAILED DESCRIPTION:
* Globally, lung cancer cases and deaths are rising. In 2018, GLOBOCAN estimated 2.09 million new cases (11.6% of total cancer cases) and 1.76 million deaths (18.4% of total cancer deaths). It is the most frequent cancer and cause of cancer death in men.
* Epidermal growth factor receptor (EGFR) mutations are the second most common oncogenic driver event in non-small cell lung cancer (NSCLC) and classical activating mutations are well defined as strong predictors for good clinical response to EGFR tyrosine kinase inhibitors (EGFRi).
* Over the last decade, the introduction of tyrosine-kinase inhibitors (TKIs) has showed a remarkable paradigm shift in the treatment of non-small cell lung cancer (NSCLC). However, genetic testing is sometimes unavailable.
* Data from previous studies that have investigated the value of F-18 FDG PET/CT for predicting EGFR status are conflicting.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC patients who underwent EGFR mutation testing.
* All patients ≥ 18 years.

Exclusion Criteria:

* Time interval between EGFR sampling and PET/CT more than 1 month.
* Patients had been treated before sampling for the gene alteration analysis
* Patients with glucose level < 200 mg/dl.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with NSCLC who are ≥ 18 years and underwent EGFR mutation testing and not treated before F-18FDG PET/CT study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
• Assessment of semi-quantitative F-18 FDG PET/CT as a non-invasive method for prediction of EGFR mutations in lung cancer patients. | baseline
  detection value of F-18 FDG PET/CT for the prediction of EGFR mutation in lung cancer patients.

SECONDARY OUTCOMES:
• Assessment of the relationship between degree of the tracer uptake and pathology of the lesion. | baseline
  correlate between degree of the tracer uptake and pathology of the lesion

REFERENCES:
- [Background] Bade BC, Dela Cruz CS. Lung Cancer 2020: Epidemiology, Etiology, and Prevention. Clin Chest Med. 2020 Mar;41(1):1-24. doi: 10.1016/j.ccm.2019.10.001. PMID 32008623
- [Background] Harrison PT, Vyse S, Huang PH. Rare epidermal growth factor receptor (EGFR) mutations in non-small cell lung cancer. Semin Cancer Biol. 2020 Apr;61:167-179. doi: 10.1016/j.semcancer.2019.09.015. Epub 2019 Sep 25. PMID 31562956
- [Background] Lv Z, Fan J, Xu J, Wu F, Huang Q, Guo M, Liao T, Liu S, Lan X, Liao S, Geng W, Jin Y. Value of 18F-FDG PET/CT for predicting EGFR mutations and positive ALK expression in patients with non-small cell lung cancer: a retrospective analysis of 849 Chinese patients. Eur J Nucl Med Mol Imaging. 2018 May;45(5):735-750. doi: 10.1007/s00259-017-3885-z. Epub 2017 Nov 21. PMID 29164298
- [Background] Huang CT, Yen RF, Cheng MF, Hsu YC, Wei PF, Tsai YJ, Tsai MF, Shih JY, Yang CH, Yang PC. Correlation of F-18 fluorodeoxyglucose-positron emission tomography maximal standardized uptake value and EGFR mutations in advanced lung adenocarcinoma. Med Oncol. 2010 Mar;27(1):9-15. doi: 10.1007/s12032-008-9160-1. Epub 2009 Jan 7. PMID 19130320